

## **Consent form**

## Effect of millet based muffins consumption on glycaemic, insulinemic response and gastric emptying in pre-diabetic adults

## **Contacts:**

Ameerah Almaski14107967@brookes.ac.ukTel: 01865 483283Dr Helen Lightowlerhlightowler@brookes.ac.ukTel: 01865 483245Dr Sangeetha Thondrepthondre@brookes.ac.ukTel: 01865 483988Dr Shelly Coescoe@brookes.ac.ukTel: 01865 483839

Functional Food Centre Department of Sport and Health Sciences Oxford Brookes University Gipsy Lane Campus Oxford OX3 0BP

| Ple | ease <u>INITIAL</u> the appropriate box | Yes | No |
|---|---|---|---|
| 1. | I confirm that I have read and understand the information sheet for the above research project. | | |
| 2. | I confirm that I have had the opportunity to ask questions and have received satisfactory answers to all my questions. | | |
| 3. | I understand that my participation is voluntary and that I am free to withdraw at any time, without giving reason, and to request for any unprocessed data previously supplied to be withdrawn. | | |
| 4. | I understand that confidentiality of information provided can only be protected within the limits of the law. | | |
| 5. | I agree to take part in the screening and the above research and give blood and breath samples | | |
| Name of Participant | | | |
| Sign | nature | | |
| Con | tact number: | | |
| ema | il: | | |
| | ne of Researcher Date | | |
| Sign | nature | | |
| Mar | ch 6 <sup>th</sup> 2017 | | |